CLINICAL TRIAL: NCT04111068
Title: Improving Vision in Adults With Macular Degeneration, Study 1: the Effect of Brain Stimulation
Brief Title: Improving Vision in Adults With Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ben Thompson, Professor; Associate Director for Research, University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VSBrainStim1
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Brain Stimulation; Psychophysics; Reading; tDCS; RSVP; Visual Acuity; Uncrowded Visual Acuity; Crowded Visual Acuity
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: 1 session of active brain stimulation and 1 session of placebo sham stimulation. Each participant will perform both sessions in a randomly-assigned order.
Who Masked: Participant, Investigator
Masking Description: The participant and the researcher will be blind to the order of the sessions for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active then Sham (Experimental): Participants in this arm will be exposed to active stimulation during session 1 and sham/placebo stimulation during session 2
  Interventions: Device: anodal tDCS Active Stimulation; Device: anodal tDCS Sham/Placebo Stimulation
- Sham then Active (Experimental): Participants in this arm will be exposed to sham/placebo stimulation during session 1 and active stimulation during session 2
  Interventions: Device: anodal tDCS Active Stimulation; Device: anodal tDCS Sham/Placebo Stimulation

INTERVENTIONS:
Device: anodal tDCS Active Stimulation — a weak electric current is applied to the head through electrodes to affect the cortical excitability of the targeted cells in the brain.
Device: anodal tDCS Sham/Placebo Stimulation — The tDCS machine will be used as in active stimulation, except the electrical current will not be applied.

SUMMARY:
The purpose of this study is to test whether a kind of brain stimulation called anodal transcranial direct current stimulation (a-tDCS) can improve the ability of people with age-related macular degeneration (AMD) or juvenile macular degeneration (JMD) to read words presented to them on a computer screen. In addition, secondary measures of visual acuity will also be examined to determine whether brain stimulation can allow patients to resolve finer details of an image. The proposed treatment is the application of a-tDCS onto the participant's head, with brain stimulation aimed at Primary Visual Cortex toward the occipital pole. The investigators will test the ability of participants to read words before and after the application of stimulation. The difference between the pre and post tests when receiving active stimulation will be compared to the difference when receiving sham stimulation, because sham stimulation is not expected to improve reading beyond a placebo. The aim of the study is to examine the potential of brain stimulation as an effective treatment for macular degeneration that may be used in conjunction with more traditional eye-based interventions. The investigators hypothesize that the brain stimulation will enable higher performance in the reading task and secondary measures due to an increase in the cortical excitability of the stimulated brain cells.

DETAILED DESCRIPTION:
This study will be carried out in Ontario, Canada (University of Waterloo) and Hong Kong (The Hong Kong Polytechnic University). There are two conditions: Active brain stimulation and sham/placebo brain stimulation. This study uses a within-subjects design, such that all participants will take part in both conditions on separate sessions.

Participants will be recruited from university-affiliated clinics and local clinical practices. Following full informed consent, participants will complete baseline testing and clinical testing to confirm that they meet eligibility criteria including: a diagnosis of macular degeneration without any additional eye disease, impaired vision but with enough visual acuity that the computer monitor can still present readable word, and no contraindications for brain stimulation interventions. Eligible participants will then be randomized to either receiving the active stimulation first or the placebo stimulation first.

The primary outcome measure is verbal reading accuracy for sentences presented on a computer screen following a Rapid Serial Visual Presentation (RSVP) task in which a single word is presented on the screen at a time. Participants will freely observe the words and will indicate the words on the screen verbally. The secondary outcome measures are crowded and uncrowded visual acuity as measured by Freiburg Visual Acuity & Contrast Test (FrACT) using the Landolt C stimulus. The "C"'s gap will be oriented randomly, and the participant will indicate the orientation of the stimulus. Crowded visual acuity will be assessed with Landolt C surrounded by a solid ring, while uncrowded visual acuity will be assessed with the Landolt C alone.

The study consists of 3 sessions:

Session 1: The first session will include the clinical evaluation. In addition, the first session will also collect the participant's individual RSVP performance threshold by presenting a variety of reading speeds and print sizes. The selected threshold will be the combination of print size and presentation speed required for a given participant to achieve roughly 55% performance accuracy.

Session 2 and 3: Brain stimulation sessions. At the start of each session, participants will perform baseline pre tests for the uncrowded and crowded visual acuity tasks as well as the RSVP task using their selected threshold from Session 1. They will then undergo a-tDCS to their primary visual cortex - this stimulation may be either active or placebo on any given day, but all participants will have been exposed to both sham and placebo by the end of Session 3. During the brain stimulation, participants will perform post tests for the primary outcome measure (RSVP) and the two secondary outcome measures (crowded and uncrowded visual acuity). Five minutes after the completion of the brain stimulation, participants will again perform all three post tests. A third set of post tests will be completed 30 minutes after the completion of the brain stimulation.

All outcome measures will be analyzed by comparing the baseline (pre test) scores to the post test scores, examining whether the active brain stimulation condition resulted in greater post test improvement relative to the placebo brain stimulation condition. The time course of the effect of brain stimulation will also be examined by comparing the effect of brain stimulation at each of the 3 post tests to one another.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AMD (age 60+) or JMD (current age 18+).
2. Central vision loss and use of a peripheral preferred retinal locus (PRL) to fixate on visual objects, as confirmed by a microperimeter.
3. Visual acuity (VA); between 0.5 and 1.0 logMAR inclusive (6/18-6/60) in the better eye.
4. Best-corrected near visual acuity of 4.0M at 40 cm or better in the better eye
5. Stable vision for the previous 3 months (by patient report).

Exclusion Criteria:

1. Diagnosed dementia.
2. Not fluent in reading English (Waterloo) or Chinese characters (Hong Kong).
3. Any ocular surgery (including anti-vegF injections) within the duration of the study.
4. Ocular pathology other than JMD or AMD that can reduce central vision.
5. Severe hearing impairment.
6. Contraindications for brain stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Rapid Serial Visual Presentation (RSVP) Reading Pre-Test | This test is roughly 6 minutes in length, occurring before brain stimulation.
  Behavioral Measure - Participants will verbally read words presented on a computer. The speed of the presentation and the size of the words will be personalized to the participant so that roughly 50% accuracy can be expected.
Rapid Serial Visual Presentation (RSVP) Reading Post-Test 1 (during stimulation) | This test is roughly 6 minutes in length, occurring during the 20 minute brain stimulation period.
  Behavioral Measure - Participants will verbally read words presented on a computer. The speed of the presentation and the size of the words will be personalized to the participant so that roughly 50% accuracy can be expected without accounting for any effects of stimulation.
Rapid Serial Visual Presentation (RSVP) Reading Post-Test 2 (5 min after stimulation) | This test is roughly 6 minutes in length, occurring 5 minutes after the completion of stimulation.
  Behavioral Measure - Participants will verbally read words presented on a computer. The speed of the presentation and the size of the words will be personalized to the participant so that roughly 50% accuracy can be expected without accounting for any effects of stimulation.
Rapid Serial Visual Presentation (RSVP) Reading Post-Test 3 (30 min after stimulation) | This test is roughly 6 minutes in length, occurring 30 minutes after the completion of stimulation.
  Behavioral Measure - Participants will verbally read words presented on a computer. The speed of the presentation and the size of the words will be personalized to the participant so that roughly 50% accuracy can be expected without accounting for any effects of stimulation.

SECONDARY OUTCOMES:
Uncrowded Visual Acuity Pre-Test | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Pre-Test" before brain stimulation.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html
Uncrowded Visual Acuity Post-Test 1 (during stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 1" while brain stimulation is ongoing.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html
Uncrowded Visual Acuity Post-Test 2 (5 min after Stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 2" 5 minutes after brain stimulation completion.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html
Uncrowded Visual Acuity Post-Test 3 (30 min after Stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 3" 30 minutes after brain stimulation completion.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html
Crowded Visual Acuity Pre-Test | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Pre-Test" before brain stimulation.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html. The Crowded Landolt C stimulus adds a solid black ring round the standard Landolt C stimulus and generally results in poorer performance.
Crowded Visual Acuity Post-Test 1 (during stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 1" while brain stimulation is ongoing.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html. The Crowded Landolt C stimulus adds a solid black ring round the standard Landolt C stimulus and generally results in poorer performance.
Crowded Visual Acuity Post-Test 2 (5 min after stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 2" 5 minutes after brain stimulation completion.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html. The Crowded Landolt C stimulus adds a solid black ring round the standard Landolt C stimulus and generally results in poorer performance.
Crowded Visual Acuity Post-Test 3 (30 min after stimulation) | Roughly 2 minutes in length, administered after the primary outcome measure "RSVP Reading Post-Test 3" 30 minutes after brain stimulation completion.
  Visual acuity as measured by participants indicating the orientation of the gap present in a Crowded Landolt C stimulus using the freely available FrACT software https://michaelbach.de/fract/index.html. The Crowded Landolt C stimulus adds a solid black ring round the standard Landolt C stimulus and generally results in poorer performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Thompson, PhD, Principal Investigator — University of Waterloo
Locations (2):
- University of Waterloo, Waterloo, Ontario, Canada
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IDP that underlie results in a publication will be available upon reasonable request to the research team.
Supporting Information: Analytic Code
Time Frame: IDP will be available upon a publication, and no more than 9 months after the publication.
Access Criteria: IDP will be shared to researchers who provide a methodologically sound proposal.

DOCUMENTS (2):
  • Study Protocol (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04111068/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT04111068/SAP_001.pdf